#### **ANNEXES AND ICF**

#### TITLE

Therapeutic exercise protocol for the prevention of anterior cruciate ligament injuries in female football players with dynamic knee valgus.

**DOCUMENT DATE:** 30/07/2023

#### **Annex I: SPIRIT checklist**

| Section/item | | Description |
|---|---|---|
| Administrative information | 4 | |
| Title | 1 | Descriptive title identifying the study design, population, interventions, and, if applicable, trial acronym |
| Trial registration | 2a | Trial identifier and registry name. If not yet registered, name of intended registry |
| | 2b | All items from the World Health Organization Trial Registration Data Set |
| Protocol version | 3 | Date and version identifier |
| Funding | 4 | Sources and types of financial, material, and other support |
| Roles and responsibilities | 5a | Names, affiliations, and roles of protocol contributors |
| | 5b | Name and contact information for the trial sponsor |
| | 5c | Role of study sponsor and funders, if any, in study design, collection, management, analysis, and interpretation of data, writing of the report; and the decision |
| | )L | submit the report for publication, including whether they will have ultimate authority over any of these activities |
| | 5d | Composition, roles, and responsibilities of the coordinating centre, steering committee, endpoint adjudication committee, data management team, and othe individuals or groups overseeing the trial, if applicable (see Item 21a for data monitoring committee) |
| Introduction | | |
| Background and rationale | 6a | Description of research question and justification for undertaking the trial, including summary of relevant studies (published and unpublished) examining benefits and harms for each intervention |
| | 6b | Explanation for choice of comparators |
| )bjectives | 7 | Specific objectives or hypotheses |
| rial design | 8 | Description of trial design including type of trial (eg, parallel group, crossover, factorial, single group), allocation ratio, and framework (eg, superiority, equivalence, noninferiority, exploratory) |
| Methods: Participants, inte | rventions | , and outcomes |
| tudy setting | 9 | Description of study settings (eg., community clinic, academic hospital) and list of countries where data will be collected. Reference to where list of study sites can be obtained |
| ligibility criteria | 10 | Inclusion and exclusion criteria for participants. If applicable, eligibility criteria for study centres and individuals who will perform the interventions (eg. |
| | | surgeons, psychotherapists) |
| nterventions | 11a | Interventions for each group with sufficient detail to allow replication, including how and when they will be administered |
| | 11b | Criteria for discontinuing or modifying allocated interventions for a given trial participant (eg, drug dose change in response to harms, participant request, or |
| | | improving/worsening disease) |
| | 110 | 7 - 0 |
| | 11c | Strategies to improve adherence to intervention protocols, and any procedures for monitoring adherence (eg, drug tablet return, laboratory tests) |
| | 11d | Relevant concomitant care and interventions that are permitted or prohibited during the trial |
| Outcomes | 12 | Primary, secondary, and other outcomes, including the specific measurement variable (eg. systolic blood pressure), analysis metric (eg. change from baselin |
| | | final value, time to event), method of aggregation (eg, median, proportion), and time point for each outcome. Explanation of the clinical relevance of chosen |
| Participant timeline | 13 | efficacy and harm outcomes is strongly recommended Time schedule of enrollment interventions (including any purple in any purple in a specific property and visits for martining and purple in the property of the property o |
| arocipani, umetine | 13 | Time schedule of enrolment, interventions (including any run-ins and washouts), assessments, and visits for participants. A schematic diagram is highly recommended (see fig 1) |
| ample size | 14 | Estimated number of participants needed to achieve study objectives and how it was determined, including clinical and statistical assumptions supporting a |
| | ** | sample size calculations |
| Recruitment | 15 | Strategies for achieving adequate participant enrolment to reach target sample size |
| Methods: Assignment of in | terventio | ns (for controlled trials) |
| llocation: | | |
| equence generation | 16a | Method of generating the allocation sequence (eg, computer-generated random numbers), and list of any factors for stratification. To reduce predictability |
| | | of a random sequence, details of any planned restriction (eg, blocking) should be provided in a separate document that is unavailable to those who enrol participants or assign interventions |
| Mocation concealment | 16b | Mechanism of implementing the allocation sequence (eg, central telephone; sequentially numbered, opaque, sealed envelopes), describing any steps to |
| nechanism | | conceal the sequence until interventions are assigned |
| | 16c | |
| mplementation | | Who will generate the allocation sequence, who will enrol participants, and who will assign participants to interventions |
| Blinding (masking) | 17a | Who will be blinded after assignment to interventions (eg. trial participants, care providers, outcome assessors, data analysts) and how |
| | 17b | If blinded, circumstances under which unblinding is permissible and procedure for revealing a participant's allocated intervention during the trial |
| Methods: Data collection, | managem | ent, and analysis |
| Data collection methods | 18a | Plans for assessment and collection of outcome, baseline, and other trial data, including any related processes to promote data quality (eg. duplicate measurements, training of assessors) and a description of study instruments (eg. questionnaires, laboratory tests) along with their reliability and validity, if |
| | | known. Reference to where data collection forms can be found, if not in the protocol |
| | 18b | Plans to promote participant retention and complete follow-up, including list of any outcome data to be collected for participants who discontinue or deviate |
| | | from intervention protocols |
| Data management | 19 | Plans for data entry, coding, security, and storage, including any related processes to promote data quality (eg, double data entry; range checks for data value |
| | | Reference to where details of data management procedures can be found, if not in the protocol |
| Statistical methods | 20a | Statistical methods for analysing primary and secondary outcomes. Reference to where other details of the statistical analysis plan can be found, if not in the |
| | | protocol |
| | 20b | Methods for any additional analyses (eg. subgroup and adjusted analyses) |
| | 20c | Definition of analysis population relating to protocol non-adherence (eg, as randomised analysis), and any statistical methods to handle missing data (eg, |
| | 200 | multiple imputation) |
| Hathada Haaliadaa | | тыперы түришкен |
| Methods: Monitoring | | |
| Data monitoring | 21a | Composition of data monitoring committee (DMC); summary of its role and reporting structure; statement of whether it is independent from the sponsor are competing interests; and reference to where further details about its charter can be found, if not in the protocol. Alternatively, an explanation of why a DMC |
| | | not needed |
| | 21b | |
| | 210 | Description of any interim analyses and stopping guidelines, including who will have access to these interim results and make the final decision to terminate the trial |
| H | 20 | |
| Harms | 22 | Plans for collecting, assessing, reporting, and managing solicited and spontaneously reported adverse events and other unintended effects of trial |
| | | interventions or trial conduct |
| Auditing | 23 | Frequency and procedures for auditing trial conduct, if any, and whether the process will be independent from investigators and the sponsor |
| Ethics and dissemination | | |
| | 24 | District the state of the state |
| Research ethics approval | 24 | Plans for seeking research ethics committee/institutional review board (REC/IRB) approval |
| Protocol amendments | 25 | Plans for communicating important protocol modifications (eg, changes to eligibility criteria, outcomes, analyses) to relevant parties (eg, investigators, REC/ |
| | | IRBs, trial participants, trial registries, journals, regulators) |
| Consent or assent | 26a | Who will obtain informed consent or assent from potential trial participants or authorised surrogates, and how (see Item 32) |
| | 26b | Additional consent provisions for collection and use of participant data and biological specimens in ancillary studies, if applicable |
| Table State | | |
| Confidentiality | 27 | How personal information about potential and enrolled participants will be collected, shared, and maintained in order to protect confidentiality before, during and affect the trial |
| | | and after the trial |
| Declaration of interests | 28 | Financial and other competing interests for principal investigators for the overall trial and each study site |
| Access to data | 29 | Statement of who will have access to the final trial dataset, and disclosure of contractual agreements that limit such access for investigators |
| Ancillary and post-trial care | 30 | Provisions, if any, for ancillary and post-trial care, and for compensation to those who suffer harm from trial participation |
| Dissemination policy | 31a | Plans for investigators and sponsor to communicate trial results to participants, healthcare professionals, the public, and other relevant groups (eg. via |
| | | publication, reporting in results databases, or other data sharing arrangements), including any publication restrictions |
| | 31b | Authorship eligibility guidelines and any intended use of professional writers |
| | | Plans, if any, for granting public access to the full protocol, participant-level dataset, and statistical code |
| | 31c | |
| Annandler | 31c | |
| informed consent materials | 32 | Model consent form and other related documentation given to participants and authorised surrogates |
| Appendices<br>Informed consent materials<br>Biological specimens | | Model consent form and other related documentation given to participants and authorised surrogates Plans for collection, laboratory evaluation, and storage of biological specimens for genetic or molecular analysis in the current trial and for future use in ancil studies, if applicable |

### Annex II: Informed consent form for study participation

| ENT | | | |
|---|---|---|---|
| NAME | [ID] | | BIRTHDATE |
| R AND DOOR) | | | PC |
| PHONE | E | EMAIL | |
| DATA OF LEGAL REPRESENTAT | IVE | BIRTH DATE | AS |
| FDDOFF | CATECORY | | |
| PROFES | SIONAL CATEGORT | | NUM. COLLEGE |
| appropriate<br>time. | | | |
| dure | I do not authorize the | performance of this p | rocedure |
| , | of | of | _ |
| | | healthcare professional | |
| | Sign | ature: | |
| DE INFORMATION AND | CONSENT | | |
| A III OIWE COOK | 7001102.11 | | |
| | of | of | |
| | | healthcare professional | |
| | Sign | ature: | |
| ation that corresponds to me<br>occess of my disease without im | | | |
| | | e my | |
| ocess of my disease without im | | | |
| ocess of my disease without im | | e my | |
| ocess of my disease without im | | of | |
| ocess of my disease without im | | ofhealthcare professional | |
| rocess of my disease without imed in the previous section. | pplying that I cannot give | ofhealthcare professional | |
| encess of my disease without imed in the previous section. | ind/or educational purp | ofhealthcare professional | |
| encess of my disease without imed in the previous section. | and/or educational purpont Authorizes: | ofhealthcare professional | |
| ed in the previous section. of ENTIFIC PURPOSES If the data used for scientific a | and/or educational purponot AUTHORIZE: Health professional: | of | |
| ed in the previous section. of ENTIFIC PURPOSES d the data used for scientific a | and/or educational purponot AUTHORIZE: Health professional: | of | |
| ed in the previous section. of ENTIFIC PURPOSES If the data used for scientific a | and/or educational purponor Authorize: Health professional: | of | |
| t | DATA OF LEGAL REPRESENTAT DATA OF LEGAL REPRESENTAT PROFES to carry out this procedure -I appropriate ime. dure , F INFORMATION ANE | PROCE NAME RAND DOOR) PHONE DATA OF LEGAL REPRESENTATIVE DNI PROFESSIONAL CATEGORY to carry out this procedure -I appropriate ime. dure I do not authorize the of Sign F INFORMATION AND CONSENT | PHONE EMAIL DATA OF LEGAL REPRESENTATIVE DNI BRITH DATE PROFESSIONAL CATEGORY to carry out this procedure -I appropriate time. dure |

In the event of non-coexistence of the spouses with shared parental authority, the father and mother must sign, otherwise the parent who holds it Personal data will be processed in accordance with Organic Law 3/2018, of December 5, Protection of Personal Data 1 and guarantee of digital rights

#### **Annex III: Timeline**



#### **Annex IV: Flow chart**



## **Annex V: Landing error system LESS**

#### LANDING ERROR SCORING SYSTEM (LESS)

| SAGGITAL VIEW: | if an error: | 02 |
|---|---|---|
| Knee Flexion Angle at Initial Contact: > 30 deg. Error if NO | 2 | 3 |
| Hip Flexion Angle at Initial Contact: Hips are Flexed Error if NO | | |
| Trunk Flexion Angle at Initial Contact: Trunk is Flexed Error if NO | | |
| 4. Knee Flexion Displacement: > 45 deg. more than Initial Contact Error if NO | | |
| 5. Hip Flexion Displacement: Hips flex more than Initial Contact Error if NO | | |
| 6. Trunk Flexion Displacement: <b>Trunk flexes more than Initial Contact Error if NO</b> | | |
| 7. Ankle Plantar-Flexion Angle at Initial Contact: Toe to heel Error if NO | | |
| FRONTAL VIEW: | | |
| 8. Initial Foot Contact: Symmetrical Error if NO | | |
| Lateral Trunk Flexion at Initial Contact: Trunk is Vertical Error if NO | | |
| 10. Knee Valgus Angle at Initial Contact: Knees over mid foot Error if NO | | |
| 11. Stance Width: < Shoulder width Error if YES | | |
| 12. Stance Width: > Shoulder width Error if YES | | |
| <ol> <li>Max IR Foot Position: Toes &gt; 30 deg. IR at max flexion<br/>Error if YES</li> </ol> | | |
| <ol> <li>Max ER Foot Position: Toes &gt; 30 deg. ER at max flexion<br/>Error if YES</li> </ol> | | |
| 15. Knee Valgus Displacement: Medial knee movement at max flexion Error if YES (Tibial tubercle inside 1 <sup>st</sup> ray) | | |
| OVERALL: | | |
| 16. Joint Displacement (Sagittal Plane) SOFT = no error, AVERAGE = 1 error, STIFF = 2 errors | | |
| 17. Overall Impression EXCELLENT = no error, AVERAGE = 1 error, POOR = 2 errors | | |
| TOTALS: | | AVG: |

#### Annex VI: SF-12 scale

I.M.P.R.E.S.S.

SF-12v2<sup>TM</sup> Health Survey
(SF-12v2 Standard, US Spanish Version 2.0)
To be completed by the PATIENT

| (For Internal Use Only) Patient Study Number | Completed By: |
|---|---|
| Visit Date (MM/DD/YY) | Visit Schedule (check appropriate box) □ Preop □ 3 mo □ 6 mo |
| /// | - □ 12 mo □ 24 mo |

| e completed by the | PATIENT | | · — — · - | 12 m | io |
|---|---|---|---|---|---|
| NSTRUCTIONS: 7 | The questions that follo | ow ask abo | ut what you th | ink about your h | ealth. |
| Your answers will le | t us know how you are | doing and to | what extent yo | ou are able to do | |
| our usual activities. | ************************************** | • | | | |
| Dlease answer each | question by checking one | hoy If yours | re not sure how | to answer | |
| | e answer what seems | | | to answer | |
| question, please | answer what seems | 3 most true | to you. | | |
| 1. In general, would | you say that your health i | s: | | | |
| | | | | 8.5 | |
| Excellent | Very good | Good | Regula | ar Bad | |
| The next assertions | s ask about activities o | r things the | t vou might de | on a normal da | v Does |
| | | | | | y. Does |
| our current health I | imit you from doing thos | e activities | or things? If so | , how much? | |
| | | | yes | Yes, | No, it |
| | | | it limits | it limits | doesn't limit |
| | | | me a lot | me a little | me much |
| 2. Moderate efforts, su | ch as moving a table, | | | | |
| | vling, or walking for more | е | | | |
| than 1 hour | 3. | | | | |
| trial Priodi | | | | | |
| 2 Olimb | | | | | |
| 3. Climb several t | loors up the stairs | | 70 - Eol | 100000000 | 0.00 |
| | ks, have you had any of the | he following | problems at wor | k or in | |
| our daily activities, du | e to your physical health? | | | | |
| | | | | | No |
| | | | | Oli | |
| 4 Did you do | less than you wanted | to? | | | |
| 4. Dia you ac | 1 1000 triair you wanted | 101 | | | |
| Did bassa ta a | ton delen sense testes si | aul. | | | |
| 경영 시간 그리고 있었다면 바다 하나 보고 있다면 사람들이 되었다. 사람들이 없었다. | top doing some tasks at | work | | | |
| or in your daily act | (IVITIES? | | | | (A) - 100 (A) |

© 1994, 2002 by QualityMetric Inc. and Medical Outcomes Trust. All Rights Reserved. SF-12™ is a registered trademark of Medical Outcomes Trust

# I.M.P.R.E.S.S. SF-12v2<sup>TM</sup> Health Survey (SF-12v2 Standard, US Spanish Version 2.0) To be completed by the PATIENT

| (For Internal Use Only) | |
|---|---|
| Patient Study Number | Completed By: |
| Visit Date (MM/DD/YY) | Visit Schedule (check appropriate box) ☐ Preop ☐ 3 mo 6 mo ☐ 12 mo 24 mo |

| nervous)? | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Yearly | ١ | lo | |
| 6. Did you do less than yo | ou would have | liked to bec | ause of | | | | | |
| an emotional probler | | | | | | L | | |
| 7. Did you not do your w<br>as carefully as usual<br>emotional? | | | | | | | | |
| 3. During the past 4 week | | | | | | | | |
| work (including work | outside the no | me and nou | senola chore | s)r | | | | |
| Nothing | A bit | Reg | ular | Quite | A | lot | | |
| een going for you in the | last 4 weeks. F | or each que | estion, answe | | | or | iv | |
| een going for you in the | last 4 weeks. F | or each que | estion, answe | | | or<br>nes eve | | Neve |
| een going for you in the<br>ow you felt. During the | last 4 weeks. F | For each que<br>s, how long. | estion, answe | r what is close | est to | | | Neve |
| een going for you in the<br>low you felt. During the<br>b. Did you feel calm and<br>peaceful? | last 4 weeks. I<br>past 4 weeks | For each que<br>s, how long. | estion, answe | r what is close | est to | | | Neve |
| eeen going for you in the low you felt. During the | last 4 weeks. I<br>past 4 weeks | For each que<br>s, how long. | estion, answe | r what is close | est to | | | Neve |
| een going for you in the<br>low you felt. During the<br>Did you feel calm and<br>peaceful? | last 4 weeks. I<br>past 4 weeks | For each que<br>s, how long. | estion, answe | r what is close | est to | | | Neve |
| een going for you in the ow you felt. During the . Did you feel calm and peaceful? | last 4 weeks. I<br>past 4 weeks | For each que<br>s, how long. | estion, answe | r what is close | est to | | | Neve |
| eeen going for you in the<br>low you felt. During the<br>b. Did you feel calm and<br>peaceful?<br>10. did you have a lot of energ<br>11. felt down and<br>sad? | last 4 weeks. If past 4 weeks | Always | Almost always | Many (trees | Sometin | | | Neve |
| 10. did you have a lot of energent of the sad? 12. During the past 4 weeks problems made it d | last 4 weeks. If past 4 weeks | Always | Almost always | Many (trees | Sometin | | | Neve |

© 1994, 2002 by QualityMetric Inc. and Medical Outcomes Trust. All Rights Reserved. SF-12™ is a registered trademark of Medical Outcomes Trust

#### Annex VII: Calculation of the sample size

| | [1] Sample sizes. Comparison of i | independent means: |
|----------|-------------------------------------|--------------------|
| Data: | | |
| | Variances: | equal |
| | Option: | Option 2 |
| | Standardized difference of means: 1 | ,000 |
| | Ratio between sample sizes: | 1.00 |
| | Confidence level: | 95.0% |
| Results: | | |

| Power (%) | | Sample size | |
|-----------|--------------|--------------|-------|
| | Population 1 | Population 2 | Total |
| 80.0 | 17 | 17 | 34 |
| 85.0 | 19 | 19 | 38 |
| 90.0 | 22 | 22 | 44 |
| 95.0 | 27 | 27 | 54 |

#### **Annex VIII: DVJ Test**



Footballers will be dropped from a box 30 cm high and immediately after landing they will perform a maximum vertical jump and hit on a force plate.

A qualitative and quantitative analysis will be carried out on the players prior to the start of the study to detect DKV and select only those who had it. This test will also be carried out on subsequent measurements to assess possible changes.

Three successful trials of all jumps executed will be recorded.

#### Qualitative analysis:

- $0 = no \ DKV$  or mid-lateral knee movement and toe alignment.
- 1 = when there is a slight DKV position of one or both knees.
- 2 = DKV in at least one knee, its alignment and that of the toes is poor and substantial amount of mean lateral movement of the knee.

#### Quantitative analysis:

The jump that gets the most points will be considered the worst jump, it will be used in the analysis and to represent the movement pattern of greatest potential risk for the player.

Each jump will be awarded one point based on the following criteria. If your feet:

- 1. leave the box or land at different times
- 2. are not parallel when landing or rotate if DKV is present
- 3. They are not separated approx. at shoulder distance
- 4. if there is any weight displacement.

**Annex IX: Programming intervention protocol** 

| SPECIFIC TRAINING PROTOCOL FOR THE PREVENTION OF ACL INJURIES | | | |
|---|---|---|---|
| 1st PHASE – ADAPTATION | 2nd PHASE – IMPROVEMENT | PHASE 3 – PERFORMANCE | EXERCISE DESCRIPTION |
| BAND WALK (3 x 1') | BAND HIP THRUST (3 x10) | SINGLE LEG HIP THRUST (3 x 10) | It consists of walking with theraband on ankles back and forth, one side and another. Progression 1: hip lift with theraband resistance Progression 2: hip lift with theraband on knees, knee extension and weight on pelvis |
| GOBLET SQUAT (3 x 10) | SQUAT (3 x 10) | SQUAT JUMP (3 x 10) | It consists of performing a squat with a weight attached to the chest. Progression 1: squat with barbell, do not lower the knees to more than 90° Progression 2: same as above + vertical jump. *In the 3 exercises a theraband will be added between the knees |

#### BOX JUMP (3 x 10)



#### DOUBLE LEG DROP JUMP (2 x 10)





#### SINGLE LEG DROP JUMP (4 x 6)\*







It consists of making a jump on a 50 cm drawer

**Progression 1**: Bounce jump + bipodal maximum vertical jump

**Progression 2**: Bounce Jump + Unipodal Maximum Vertical Jump

\*2 sets with each leg

#### SQUAT JUMPS (3 x 10)





#### 90° VERTICAL JUMP (3 x 10)





#### 180° JUMPS (3 x 10)





It consists of making a jump and landing in the same place going down to squat.

**Progression 1**: Jump and make a 90° turn

**Progression 2:** Jump and make a 180° turn

#### BAND LUNGE (3 x 10)



#### WEIGHT BAND LUNGE (3 x 10)



#### JUMP LUNGE (SCISSOR JUMPS) (3 x 10)





It consists of making an anterior stride, at 45° and 90° (several directions) with theraband.

**Progression 1**: multi-direction stride + chest weight + theraband to stabilize knee

**Progression 2**: Dynamic strides with weight

STIFF LEG DEADLIFT + BALL GLUTE BRIDGE BOTH KNEES (3 x 10)







SINGLE LEG DEADLIFT + BALL GLUTE BRIDGE ONE KNEE (3 x10)





#### NORDIC HAMSTRINGS (2 x 8)\*



It consists of performing 1st and 3rd series of deadlift with weight and the 2nd gluteal bridge on bipodal fitball performing flexoextension knees

**Progression 1**: deadlift with weight and gluteal bridge on unipodal flex-knee extension fitball

**Progression 2**: hamstring eccentric.

\*1st series with straight body and 2nd series with inclined body. When it passes 45° drop slowly.

#### PLANK + SIDE PLANCK (4 x 30')





PLANK TO PRESS + PLANK KNEE TO CHEST + PELVIC RETROVERSION AND ANTEVERSION + SIDE PLANK WITH HIP ABDUCTION (4 x 30')









#### SWISS BALL PLANK (6 x 10)





It consists of making 2 series of plate in prone position and 2 in lateral decubitus position.

Progression 1: 1st series plate with elbow-hand support + 2nd series knees to the chest + 3rd retro series and pelvic anteversion + 4th series side plate with hip abduction

**Progression 2**: 3 sets with elbows on fitball (flex-ext + circles) and 3 sets feet on fitball (flex-ext knees)

#### BULGARIAN SPLIT SQUAT (3 x 10)



CROSSOVER HOP-STICK (3 x 10)



#### SINGLE LEG CROSSOVER DROP (4 x 6)



It consists of making a stride and keeping the leg behind on a surface

**Progression 1**: unipodal zig-zag jumps

**Progression 2:** unipodal cross fall from 50 cm drawer. 2 series with right leg support and 2 others with left leg support

#### BOSU BOTH KNEES DEEP HOLD-MEDICINE BALL CATCH (3 x 30')



## BOSU BOTH KNEES DEEP HOLD – KICK BALL (3 x 30')



# LATERAL SQUAT JUMPS OVER THE BOSU (3 x 30')



It consists of maintaining bipodal balance on BOSU while throwing a soccer ball.

**Progression 1**: keep balance on BOSU unipodal + ball kick with inside leg or head shot

**Progression 2**: unipodal lateral jump with support on BOSU

RUSSIAN TWIST + CRUNCHES (6 x 25)



DOUBLE CRUNCHES (6 x 25)



ABDOMINAL ROLLER (4 x 10)



It consists of performing 3 sets of abdominals with trunk turns + soccer ball and another 3 series of conventional abdominals

**Progression 1**: abs with knee flexion + medicine ball between knees

**Progression 2**: eccentric abdominal exercise with abdominal roller

<sup>\*</sup>In all exercises with weight, you will work with loads between 70-80% of 1RM

<sup>\*</sup> The height of the drawer of the exercises that is required will increase depending on the progression of the athletes, starting with a drawer of 50 cm in height *Photographs taken of a CF Monnegre Mutxamel player, who gave her consent to appear in the photos without pixelating her face* 

Annex X: Infographic action protocol for women's football coaches

